CLINICAL TRIAL: NCT02890056
Title: A Culturally-tailored Narrative Intervention to Target Disparities in Obesity
Brief Title: A Community-based Study to Target Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Monica Li-Sha Wang, Assistant Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-34445; 1K01DK102447 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: sugar-sweetened beverage consumption; water consumption; dietary behaviors; youth
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H2GO! intervention (Experimental): H2GO! is a community-based behavioral intervention to reduce sugar-sweetened beverage consumption and promote water intake among school-age youth and parents.The intervention consists of 6 weekly group-based sessions (1-hour sessions twice a week) that target beverage knowledge, attitudes, and behaviors through interactive activities, youth-produced narratives, and parent-child activities. The intervention is delivered through a youth-based community setting (Boys and Girls Clubs of America) by trained Boys and Girls Club staff.
  Interventions: Behavioral: H2GO!
- Comparison (No Intervention): Usual care will take place at the comparison site (standard programming at the Boys and Girls Club comparison site).

INTERVENTIONS:
Behavioral: H2GO!
  Arms: H2GO! intervention

SUMMARY:
The purpose of this study is to determine the efficacy of a community-based behavioral intervention (H2GO!) on decreasing sugar-sweetened beverage consumption and promoting water consumption among school-aged youth and parents/caregivers. We hypothesize that participants in the intervention site will demonstrate reduced sugar-sweetened beverage intake intake and increased water intake compared to participants in the comparison site at 2 and 6 months follow-up.

DETAILED DESCRIPTION:
This study aims to assess the efficacy of a community-based behavioral intervention (H2GO!) targeting sugar-sweetened beverage and water consumption among 108 parent-child pairs (N=216) through a site-randomized trial.

The study setting includes 2 Boys and Girls Club sites in Massachusetts, USA that were pair-matched for size and racial/ethnic composition. The Boys and Girls of America is a national organization that provides affordable after-school programs for a large population (~4 million annually) of diverse youth (33% White, 30% Black, 23% Latino) from predominantly low socioeconomic backgrounds through over 4,000 club facilities across the U.S.

The H2GO! intervention was designed to address two behavioral targets: reducing the number of sugar-sweetened beverage servings consumed per day (recommended guideline of zero servings per day) and promoting water consumption (approximately 5-8 cups per day for youth participants and 8 cups per day for parental participants). Informed by the Social Cognitive Theory and the Social Ecological Model, the H2GO! Intervention was designed to target child and parent participants' knowledge, attitudes (self-efficacy, outcome expectations, perceived social norms) and behavioral capabilities related to sugar-sweetened beverage and water consumption.

The 6-week behavioral intervention consists of group-based weekly sessions (1-hour sessions twice a week) delivered by trained Boys and Girls Club program staff at the Boys and Girls Club site. Each intervention session consists of a 1-hour health module followed by a 1-hour narrative module. Topics of the health modules include: understanding the benefits of water, sampling different types of fruit-flavored water, identifying sugar-sweetened beverages, exploring the local grocery store, identifying barriers and facilitators to drinking water, and managing triggers for sugar-sweetened beverages. The narrative modules include intervention objectives and activities that reinforce knowledge, attitudes, skills, and behaviors targeted in the previous health component.

Child participants will receive a reusable water bottle and a pictorial intervention booklet. Developed by the study principal investigator (PI) and research assistants, the brightly-colored booklet was culturally and linguistically-tailored to the study population and included intervention activity worksheets, parent-child take-home activities, fun facts and quizzes, and beverage consumption tracking sheets. Activity worksheets will be completed by participants during intervention sessions; and parent-child take-home activities will be completed following each session.

Study assessments will take place at baseline, 2 months, and 6 months.

ELIGIBILITY:
This study recruits parent/caregiver-child pairs. The inclusion and exclusion criteria are further specified based on parent/caregiver participants and child participants.

Child Inclusion Criteria:

* ages 9-12 years
* current member at the Boys and Girls Club study site
* able to understand and communicate in English
* able and willing to provide consent
* parental/caregiver permission to participate

Child Exclusion Criteria:

- medical condition that limits ability to change beverage consumption behaviors

Parent/Caregiver Inclusion Criteria:

* ages 18+ years
* parent/caregiver to a Boys and Girls Club child member
* able to understand and communicate in English
* able and willing to provide consent

Parent/Caregiver Exclusion Criteria:

- medical condition that limits ability to change beverage consumption behaviors

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sugar-sweetened beverage consumption | Change from baseline to 6 months
  Measured through self-report survey
Water consumption | Change from baseline to 6 months
  Measured through self-report survey

SECONDARY OUTCOMES:
Body mass index percentile (age- and sex-specific) | Change from baseline to 6 months
  Trained staff will obtain child participants' height (inches) and weight (pounds) using standardized equipment. Height and weight will then be used to calculate body mass index (kg/m^2). Body mass index percentiles will be calculated using age- and sex-specific body mass index-based growth trajectories.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Wang, ScD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Pblic Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang ML, Otis M, Rosal MC, Griecci CF, Lemon SC. Reducing sugary drink intake through youth empowerment: results from a pilot-site randomized study. Int J Behav Nutr Phys Act. 2019 Jul 30;16(1):58. doi: 10.1186/s12966-019-0819-0. PMID 31362753
- [Derived] Wang ML, Lemon SC, Clausen K, Whyte J, Rosal MC. Design and methods for a community-based intervention to reduce sugar-sweetened beverage consumption among youth: H2GO! study. BMC Public Health. 2016 Nov 9;16(1):1150. doi: 10.1186/s12889-016-3803-5. PMID 27829397